CLINICAL TRIAL: NCT06982950
Title: Longitudinal Reciprocal Relationships Between Cannabis Use, Sleep, and the HPA-axis (CaSS)
Brief Title: Cannabis Association With Sleep Study
Acronym: CaSS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Nicole Bowles, Assitant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB28366
Record Dates: First submitted 2025-05-03; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Sleep
Keywords: Sleep, slow wave; Polysomnography; Marijuana Abuse; Cannabinoids; Ecological Momentary Assessment; Sleep Duration
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Intervention Model Description: After a baseline assessment of sleep, participants will undergo either 2 nights of restricted sleep (4h time in bed [TIB]) followed by a recovery sleep, OR 3 nights of an extended sleep opportunity (10h TIB)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Restriction (Experimental): After a baseline assessment of sleep, participants in this arm will undergo 2 nights of restricted sleep (4 hour time in bed).
  Interventions: Other: Manipulation of Sleep Duration
- Sleep Extension (Experimental): After a baseline assessment of sleep, participants in this arm will undergo 3 nights of an extended sleep opportunity (10 hour time in bed).
  Interventions: Other: Manipulation of Sleep Duration

INTERVENTIONS:
Other: Manipulation of Sleep Duration — After a baseline assessment of sleep, participants will undergo either 2 nights of restricted sleep (4 hour time in bed) followed by a recovery sleep, OR 3 nights of an extended sleep opportunity (10 hour time in bed)

SUMMARY:
The purpose of this study is to learn more about cannabis use, sleep, and stress, and whether there is any relationship between the three.

DETAILED DESCRIPTION:
After passing a physical assessment and psychological screen, 60 participants will be enrolled. Ahead of the 21-day protocol participants will report to our laboratory sleep facilities and will be set-up to perform a full polysomnography test (monitored overnight sleep with equipment including superficial electrodes, heart rate [HR] monitor, breathing monitors). This initial night of sleep with study equipment is provided in order to reduce sleep differences based on sleeping in a new environment and the burden of wearing equipment while sleeping. Before and after this 8h sleep period participants will be introduced to all surveys and behavioral testing that will be used as part of the experimental nights. Participants who complete the familiarization night will be randomized to two different possible experimental protocols that differ in the length of the sleep period. In order to fully characterize cannabis use behaviors (frequency, amount, mode of use) on sleep in an individual's typical environment (i.e. in the places and during the activities of normal living), we will implement 21 days of activity monitoring via multiple daily surveys (which collectively is a research strategy known as Ecological Monitoring Assessment [i.e., EMA]) along with concurrent actigraphy, that is, the monitoring of movement via the use of a wrist-worn watch-like device. Approximately one-week into this observational period, participants will complete the 2 x 4-night experimental nights (consecutive nights) with a washout (return to habitual sleep patterns) of at least 6 days.

Participants are able to spend the day outside of the laboratory during the experimental night period (i.e. they will come into the lab each night to sleep, and have their sleep monitored, but able to do normal activities during the days). Following in laboratory assessments, participants will complete any remaining at home assessments needed for 21 days of EMA/actigraphy.

ELIGIBILITY:
Inclusion Criteria:

* fluent in English
* 18.5<BMI<40 kg/m2
* no shift work in the last 12 months
* no travel across time zones in the last 2 months.

Exclusion Criteria:

* Chronic disease-Medical history/prior diagnosis of the following:
* cardiometabolic disease (e.g., myocardial infarction, angina, diabetes)
* essential hypertension
* hepatic impairment
* severe obstructive sleep apnea
* restless legs syndrome
* parasomnia
* neurological disease (e.g., early onset dementia)
* unstable psychiatric disorders (e.g., bipolar disorder, schizophrenia, major depression with suicidality).
* Drug/Alcohol use criteria:
* Illicit drugs apart from cannabis or related products are prohibitive.
* Volunteers may consume caffeine, however, >3 cups of coffee (or otherwise equivalent of >300mg/day) is prohibitive.
* Participants who consume >14 alcoholic drinks/week and/or have a diagnosis (or history) of alcohol use disorder will be excluded (a toxicological urine screen will be conducted to verify reported non-use during the initial screening and on the day of admission to the in-laboratory portion of the study).
* Use of prescription or over-the-counter medications or supplements that affect sleep are also exclusionary.
* Contraceptives are required for women and will continue to be taken throughout the experiment.
* Prior Shift Work:
* Volunteers must have no history of working irregular day and night hours, regular night work, or rotating shift work for the 3 months prior to the study.

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2032-06-30 (Estimated)

PRIMARY OUTCOMES:
Daily Cannabis Use Frequency | Assessed in surveys performed 4 times per day, and across the entire 21-day study
  The number of smoking/vaping sessions per day.
Wake After Sleep Onset (WASO) | 21 days
  Wake after sleep onset (measured in minutes) will be assessed each night from actigraphy; larger value indicates greater disruptions to sleep.
Cortisol Awakening Response | 8 nights
  Salivary cortisol levels assessed as the difference between waking and peak levels assessed ~30-45 minutes after awakening.

SECONDARY OUTCOMES:
Wake After Sleep Onset (Polysomnography) | 8 nights
  Wake after sleep onset (measured in minutes) will be assessed each night of the in laboratory study using polysomnography [PSG]); larger value indicates greater disruptions to sleep.
Sleep Latency | 8 nights
  Measured in minutes and assessed each night of the in laboratory study using polysomnography; assessed at time from in bed and lights off to any stage of sleep including Non rapid eye movement (NREM) 1.
Total Sleep Time | up to 21 days
  Measured (in minutes)from actigraphy (21 days of data) and in laboratory study using polysomnography (8 nights of data).
Sleep Macroarchitecture | 8 nights
  Non rapid eye movement (NREM) 1-3 and Rapid eye movement (REM), time and %, assessed each night of the in laboratory study using polysomnography.
Sleep Microarchitecture | 8 nights
  Delta power, theta power, and alpha power during quiet wakefulness and sleep assessed during the in laboratory study using polysomnography.
Median Reaction Time | 8 days
  Assessed from a 10 minute psychomotor vigilance test approximately hourly during the in laboratory component of the study; larger value indicates reduced vigilance.
Time to NREM1 Sleep (modified Maintenance of Wakefulness) | 8 days
  Assessment of sleep pressure using a modified Maintenance of Wakefulness test provided approximately hourly during the in laboratory component of the study.
Subjective Sleepiness | 21 days
  Assessed 4-5 times/day as part of the Ecological Monitoring Assessment (EMA) and approximately hourly during the in laboratory component of the study using the Karolinska Sleepiness Scale (KSS). The KSS uses a 9-point scale with 1 = extremely alert and 9 = extremely sleepy - fighting sleep.
Pre-Ejection Period | 8 days
  Using continuous electrocardiogram (EKG) during the in laboratory portion of the study we will calculate the interval between the Q wave on the EKG signal and the B point on the dZ/dt signal.
Sleep High Frequency Heart Rate Variability (HRV) | 8 nights
  Assessed from continuous EKG during the in laboratory portion of the study, high frequency (HF; 0.15-0.4 Hz) HRV will be calculated by passing R-R intervals through a fast Fourier power spectral analysis on all 2-minute periods of nocturnal EKG of stable PSG identified sleep.
Mood | 21 days
  Daily assessments of mood will be collected during the EMA using abbreviated versions of Profile of Mood States (POMS) with each mood description rated on a 5-point scale between not at all (0) to extremely (4).
Cannabis Use Composite Score | 21 days
  Composite score based on daily frequency of use, amount of use, time of use, and method of use.
Positive Affect | 21 days
  Daily assessments of positive affect will be collected during the EMA using The Positive and Negative Affect Schedule (PANAS) scales with values ranging from 10-50 (high score representing higher levels of positive affect).
Negative Affect | 21 days
  Daily assessments of negative affect will be collected during the EMA using the PANAS with values ranging from 10-50 (lower scores representing lower levels of negative affect).
Sleep Low Frequency HRV | 8 nights
  Assessed from continuous EKG during the in laboratory portion of the study, low frequency (LF; 0.04-0.15 Hz) HRV will be calculated by passing R-R intervals through a fast Fourier power spectral analysis on all 2-minute periods of nocturnal EKG of stable PSG identified sleep.
Sleep Normalized HF Power | 8 nights
  Normalized HF power is calculated by dividing integrated HF spectra by the total power (LF+HF) and multiplying by 100.
Sleep standard deviation of the R-R interval of normal sinus beats (SDNN) | 8 nights
  Time domain HRV will be expressed using the standard deviation of the R-R interval of normal sinus beats (SDNN) during stable 2-minute segments of sleep.
Area under the curve of the CAR | 8 nights
  Total amount of cortisol secreted after awakening assessed using the trapezoidal rule to assess area under the curve from waking to 60 minutes post waking saliva cortisol levels.

IPD SHARING:
Plan to Share IPD: Yes